CLINICAL TRIAL: NCT01404520
Title: Patient Activation, Counseling and Exercise - Acute Leukemia (PACE-AL) Health Promoting Rehabilitation. A Multimodal Exercise-based Intervention in Patients With Acute Leukaemia Undergoing Re-induction or Consolidation Chemotherapy
Brief Title: Patient Activation, Counseling and Exercise - Acute Leukemia (PACE-AL)
Acronym: PACE-AL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitetshospitalernes Center for Sygepleje (Other)
Collaborators: University of Copenhagen (Other); Novo Nordisk A/S (Industry); Danish Cancer Society (Other); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Mary Jarden, Research Fellow, Universitetshospitalernes Center for Sygepleje
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-4-2010-046
Record Dates: First submitted 2011-05-10; First posted 2011-07-28 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Acute Leukemia
Keywords: #14 Cancer Related fatigue; #13 Quality of Life; #12 "Psychosocial Intervention"[ti/ab]; #11 Rehabilitation[tw]; #10 "Physical Fitness"[tw]; #9 "Physical Activity"[tw]; #8 "Exercise Therapy"[tw]; #7 Exercise[tw]; #6 Hematologic[tw]; #5 Hematological[tw]; #4 Leukemia, Myeloid, Acute[mh]; #3 "Acute Myeloid Leukemia"[tw]; #2 "Acute Lymphoblastic Leukemia"[tw]; #1 "Acute Leukemia"[tw]

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise based multimodal intervention (Experimental): The intervention is initiated early, during treatment (consolidation) in the intra-hospital setting and continues for two successive treatment series (12 weeks). The intervention is a three hour/wk supervised in-hospital programme of aerobic (stationary cycle) and functional muscle training, progressive relaxation training, nutrition supplement (protein and carbohydrate) immediately after training and health-promoting consultation combined with an unsupervised in-home walking and progressive relaxation programme
  Interventions: Other: Exercise based multimodal intervention
- Control Group (No Intervention): Control group receives usual care

INTERVENTIONS:
Other: Exercise based multimodal intervention — The intervention is initiated early, during treatment (consolidation) in the intra-hospital setting and continues for two successive treatment series (12 weeks). The intervention is a three hour/wk supervised in-hospital programme of aerobic (stationary cycle) and functional muscle training, progressive relaxation training, nutrition supplement (protein and carbohydrate) immediately after training and health-promoting consultation combined with an unsupervised in-home walking and progressive relaxation programme.
  Arms: Exercise based multimodal intervention

SUMMARY:
The purpose of this study is to test a new preventive and restorative intervention for patients with acute leukaemia undergoing consolidation chemotherapy, to measure and delineate the patients' treatment related symptom burden and to explore the effect of the intervention on length of hospital stay, duration of sick leave and return to work status. Further, to examine the relationship of the symptom profile with clinical indicators, physiological response, physical performance and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are able to speak Danish > 18 years and newly diagnosed with acute leukæmia (MDS, AML, CMML, APL or ALL)
* Normal EKG, blood pressure and pulse
* Signed informed written consent

Exclusion Criteria:

* Medical reason that contraindicates physical activity
* Patients diagnosed with a symptomatic cardial disease
* Documented bone metastasis
* Cognitively or emotionally unstable
* Unable to read or write in Danish
* Patients unable to carry out baseline tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Distance 6MWD | Change from baseline in 6MWD at 12 weeks
  Change in distance in meter

SECONDARY OUTCOMES:
Estimated VO2 max Aastrand test | Change from baseline in VO2 Aastrand test at 12 weeks
  Change in l/m
Timed chair stand | Change from baseline in timed chair stand at 12 weeks
  Change in number of repetitions
Timed biceps curl | Change from baseline in timed bicep curl at 12 weeks
  Change in number of repetitions
EORTC QLQ-C30 | Change from baseline in EORTC QLQ-C30 at 12 weeks
  Change in scores for quality of life
FACT-An | Change from baseline in FACT-An at 12 weeks
  Change in scores for quality of life/function
HADS | Change from baseline in HADS at 12 weeks
  Change in scores for emotional wellbeing
SF36 | Change from baseline in SF36 at 12 weeks
  Change in scores for general health
MDASI | Change from baseline over time (1,2,3,4,5,6,7,8,9,10,11,12 weeks)
  Change in scores for symptom burden

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jarden, Ph.D., Principal Investigator — UCSF and CIRE
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital Rigshospital, Copenhagen
  - Herlev Hospital, Herlev

REFERENCES:
- [Derived] Jarden M, Moller T, Christensen KB, Kjeldsen L, Birgens HS, Adamsen L. Multimodal intervention integrated into the clinical management of acute leukemia improves physical function and quality of life during consolidation chemotherapy: a randomized trial 'PACE-AL'. Haematologica. 2016 Jul;101(7):e316-9. doi: 10.3324/haematol.2015.140152. Epub 2016 Apr 1. No abstract available. PMID 27036163
- [Derived] Jarden M, Moller T, Kjeldsen L, Birgens H, Christensen JF, Bang Christensen K, Diderichsen F, Hendriksen C, Adamsen L. Patient Activation through Counseling and Exercise--Acute Leukemia (PACE-AL)--a randomized controlled trial. BMC Cancer. 2013 Oct 2;13:446. doi: 10.1186/1471-2407-13-446. PMID 24083543